CLINICAL TRIAL: NCT00319566
Title: Heart and Estrogen-Progestin Replacement Study (HERS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: 713B-401-US
Record Dates: First submitted 2006-04-27; First posted 2006-04-27 (Estimated); Last update posted 2006-04-27 (Estimated); Status verified 2002-01

CONDITIONS: Coronary Heart Disease
Keywords: Coronary Heart Disease; Hormone replacement therapy; Estrogen; Postmenopausal women
MeSH Terms: conditions — Coronary Disease | interventions — Estrogens, Conjugated (USP); Medroxyprogesterone

INTERVENTIONS:
Drug: Premarin .625 mg daily plus medroxyprogesterone 2.5 mg daily

SUMMARY:
The purpose of the study is to determine whether hormone replacement therapy in post menopausal women with coronary artery disease prevents future heart attacks or death from coronary heart disease.

DETAILED DESCRIPTION:
A randomized, blinded trial in post menopausal women with cornaornary artery disease to test the hypothesis, among 2340 women who have a uterus, that those randomized to receive estrogen-progestin replacement therapy (Premanrin .625 mg daily plus medroxygrprogesterone acetate 2.5 mg daily) have the same frequency on new CHD events (myocardial infarction and CHD death) as those randomized to placebo.

ELIGIBILITY:
Inclusion Criteria:

* <75 y.o.
* uterus present
* postmenopausal
* evidence of CHD
* signed consent

Exclusion Criteria:

* MI, CABG, mechanical revascularization within 6 months
* serum triglyceride >300mg/dl
* used hormone therapy or estrogen vaginal cream in past 3 months
* history of DVT or pulmonary embolism
* history of breast cancer or mammogram suggestive of cancer
* history of endometrial cancer
* abnormal uterine bleeding
* pap smear abnormal
* SGOT more than 1.2 times normal
* Disease judged to be fatal within 4 yrs
* alcoholism, drug abuse
* NYHA Class IV congestive heart failure
* uncontrolled hypertension
* uncontrolled diabetes
* participation in any other investigational study

Ages: 55 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2430
Dates: Start 1992-07; Study Completion 2001-07

PRIMARY OUTCOMES:
Myocardial Infarction
CHD Death

SECONDARY OUTCOMES:
CABG, revascularization, angina
serum lipids
quality of life
compliance
incidence of uterine bleeding and endometrial hyperplasia
incidencet and severity of vasomotor and genitourinary symptoms
adverse effects
thromboembolic events
symptomatic gallbladder disease
fractures
cancer
stroke
peripheral arterial disease
total mortality

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Hulley, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States